CLINICAL TRIAL: NCT01661413
Title: Chemotherapy-induced Nausea and Vomiting in Children Receiving Intrathecal Methotrexate With/Without Vincristine
Brief Title: Nausea and Vomiting in Children Receiving Chemotherapeautic Monotherapy
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Angela Punnett, Staff Physician, The Hospital for Sick Children
Other Study IDs: 1000030743
Record Dates: First submitted 2012-08-07; First posted 2012-08-09 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Acute Leukemia
Keywords: Acute Leukemia; Pediatrics; Intrathecal methotrexate; Chemotherapy; Nausea; Vomiting
MeSH Terms: conditions — Nausea; Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute Leukemia: Children diagnosed with acute leukemia, undergoing chemotherapy. Patients with acute leukemia will receive intrathecal methotrexate on day 1 plus intravenous vincristine on day 1 plus oral steroid on days 1-5 plus their regularly scheduled and ongoing daily oral 6-mercaptopurine at the start of a maintenance therapy cycle.

SUMMARY:
Chemotherapy induced nausea is a common side effect for children undergoing chemotherapy. Furthermore, chemotherapy-induced vomiting is a major factor limiting quality of life during treatment reported by paediatric cancer survivors. Complete prevention of both nausea and vomiting is the goal of anti-vomiting and nausea medications. It is important to understand whether or not certain chemotherapeutic treatments are more or less likely to cause these symptoms. Acute leukemia is the most common cancer diagnosed in children. Intrathecal methotrexate is an important part of chemotherapy for the prevention and treatment of central nervous system leukemia over the 2.5 to 3.5 years of the treatment program for leukemia. The likelihood that intrathecal methotrexate administered as monotherapy will cause nausea and vomiting has not yet been described in children. Knowledge of the likelihood that intrathecal methotrexate will cause nausea and vomiting will therefore be important to optimize treatment for these side-effects of chemotherapy. The primary aim of this prospective study is to evaluate the potential of intrathecal methotrexate to cause nausea and vomiting in paediatric cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* 4 years old to 18 years of age (age range in which the PeNAT has been validated) [18]
* English speaking (PeNAT has been validated only in English)
* Cognitive ability of the child believed to be at least at a 4 year old level according to parent or health care professional
* Patients are past their first cycle of maintenance therapy to avoid interactions with the intensive chemotherapy phase.

Exclusion Criteria:

* Receiving chemotherapy other than dictated by protocol for maintenance therapy within 24 hours prior to or 24 hours following receipt of intrathecal methotrexate

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Receiving intrathecal methotrexate in the context of maintenance therapy for acute lymphoblastic leukemia and as dosed by age per protocol. Patients will also receive their protocol driven maintenance chemotherapy which includes oral 6 mercaptopurine and may include IV vincristine and an oral steroid pulse (prednisone or dexamethasone). Oral methotrexate is typically held the weeks that patients receive intrathecal methotrexate during maintenance therapy.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2012-05-07 (Actual); Primary Completion 2015-10-31 (Actual); Study Completion 2015-10-31 (Actual)

PRIMARY OUTCOMES:
Acute Chemotherapy-Induced Nausea and Vomiting | Over 24 hours after receiving intrathecal methotrexate on day 1
  To describe the prevalence of acute phase CINV in these patients. Acute CINV is defined as nausea, vomiting or retching occurring within the first 24 hours following chemotherapy.

SECONDARY OUTCOMES:
Anticipatory Chemotherapy-Induced Nausea and Vomiting | Baseline
  To describe the prevalence of anticipatory nausea and vomiting in these patients. Anticipatorty nausea and vomiting begins prior to the administration of chemotherapy in patients who have previously received chemotherapy.
Delayed Chemotherapy-Induced Nausea and Vomiting | Over 168 hours (7 days) after receiving first treatment of intrathecal methotrexate
  To describe the prevalence of delayed phase CINV in these patients. Delayed CINV develops after the initial 24 hours and might last up to 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Punnett, MD, Principal Investigator — The Hospital for Sick Children; Lee Dupuis, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada